CLINICAL TRIAL: NCT05547282
Title: A Clinical Study of Low-dose Radiotherapy Combined With Conventional Radiotherapy in Patients With Malignant Tumors After Immunotherapy Failure
Brief Title: Low-dose Radiotherapy Combined With Conventional Radiotherapy After Immunotherapy Failure
Acronym: FL001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiandong Zhang (Other)
Responsible Party: Sponsor-Investigator, Jiandong Zhang, Chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(074)
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cancer Patients
Keywords: Cancer patients after immunotherapy failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose radiotherapy combined with conventional radiotherapy after immunotherapy failure (Other): The chest, abdomen and pelvis were located by enhanced CT, and the target area was delineated. The lesions were visible lymph nodes with short diameter ≥1cm, and there were metastases confirmed by two associate chief physicians by enhanced MR and PET/CT examination results.
  The primary lesion, the largest metastatic lesion or the lesion causing symptoms were selected and divided into 1.8-2Gy/F,40Gy-60Gy. For the remaining lesions, at least one easily evaluated and measurable lesion was selected as the observation lesion, and the unselected lesions (≤10 lesions) were given 1.6Gy/f, 1f/w, 4-6 times.
  Immunotherapy regimens are administered according to the specific dose and interval of the original immunization regimen, such as concurrent chemotherapy or antiangiogenic drug therapy regimens. He used Nivolumab, Pembrolizumab, Troripalimab and Camrelizumanb.
  Immunotherapy was performed at a frequency of 3 weeks in combination with radiotherapy until progression.
  Interventions: Radiation: At the same time, the original regimen of immunomaintenance therapy was continued, according to the frequency of the original immunization regimen once every 3 weeks until progress.

INTERVENTIONS:
Radiation: At the same time, the original regimen of immunomaintenance therapy was continued, according to the frequency of the original immunization regimen once every 3 weeks until progress. — At the same time, the original regimen of immunomaintenance therapy was continued, according to the frequency of the original immunization regimen once every 3 weeks until progress.

SUMMARY:
Response was evaluated according to the Guidelines for Response Criteria for Use in Trials Testing Immunotherapeutics (iRECIST) : ORR-To evaluate the objective effective rate of LDRT combined with SFRT and immunotherapy in patients with malignant tumors after immunotherapy resistance without standard regimens. PFS-To evaluate the progression-free survival (PFS) of patients with advanced malignant tumors after LDRT combined with SFRT and immunotherapy without standard regimens after immunotherapy resistance.DCR-To evaluate the proportion of patients with optimal response to LDRT and SFRT combined with immunotherapy to achieve complete response, partial response, or disease control after no standard regimen was available for immunotherapy resistance.HRQoL, AE and sAE-Evaluation of health related quality of life and safety of post-LDRT combined with SFRT and immunotherapy in patients with malignant tumors. To evaluate the benefit of patients in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient understood, participated voluntarily and signed the informed consent

  2. Age 18-65

  3. Cytologically or histologically confirmed malignancy

  4. Complete clinical data

  5. The number of primary and regional metastatic lymph nodes and distant metastatic lesions was ≤10, and the number of organ metastases was ≤5.

  6. Patients with malignant tumors who are resistant to immunotherapy (the patient's disease progression is evaluated after 6-8 weeks of treatment without improvement of clinical symptoms), and no standard treatment options are available.

  7. Measurable primary lesions and regions

Exclusion Criteria:

* 1. Missing key patient data

  2. Refusing or not cooperating with the study

  3. Patients who have participated in other clinical studies/trials within 3 months

  4. Patients with brain metastases

  5. Patients with any conditions that the investigator judged to be ineligible for study participation

  6. Patients with uncontrolled severe medical diseases who cannot tolerate radiotherapy

  7. Past immune-related side effects (immune myocarditis, pneumonia, etc.)

  8. Previous history of radiation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Eighteen months
  To evaluate the objective effective rate of LDRT combined with SFRT and immunotherapy in patients with malignant tumors after immunotherapy resistance without standard regimens.

SECONDARY OUTCOMES:
PFS | Eighteen months
  To evaluate the progression-free survival (PFS) of patients with advanced malignant tumors after LDRT combined with SFRT and immunotherapy without standard regimens after immunotherapy resistance.
DCR | Eighteen months
  To evaluate the proportion of patients with optimal response to LDRT and SFRT combined with immunotherapy to achieve complete response, partial response, or disease control after no standard regimen was available for immunotherapy resistance.
HRQoL、AE、SAE | Eighteen months
  Evaluation of health related quality of life and safety of post-LDRT combined with SFRT and immunotherapy in patients with malignant tumors.

CONTACTS AND LOCATIONS:
Overall Officials: PINGPING HU HU, Dr, Principal Investigator — Deputy chief physician
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital)16766 Jingshi Road, Jinan City, Jinan, In Shandong Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bates JE, Morris CG, Milano MT, Yeung AR, Hoppe BS. Immunotherapy with hypofractionated radiotherapy in metastatic non-small cell lung cancer: An analysis of the National Cancer Database. Radiother Oncol. 2019 Sep;138:75-79. doi: 10.1016/j.radonc.2019.06.004. Epub 2019 Jun 25. PMID 31252297